CLINICAL TRIAL: NCT03138070
Title: A Window of Opportunity Study to Assess the Modulation of Biomarkers in Head and Neck Squamous Cell Cancer (HNSCC) By Preoperative Treatment With BYL719
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Window of Opportunity
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Squamous Cell Cancer
MeSH Terms: interventions — Alpelisib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): 14 days of BYL719 treatment, open label
  Interventions: Drug: BYL719

INTERVENTIONS:
Drug: BYL719 — BYL719 400 mg daily by mouth continue for 14 days
  Other Names: Alpelisib

SUMMARY:
Single centre, single arm, preoperative window of opportunity study with a biomarker endpoint (expression profiling by RNA sequencing). Patients with resectable, histologically confirmed head and neck squamous cell carcinoma (HNSCC) for whom surgical treatment is planned as definitive management will be eligible.

DETAILED DESCRIPTION:
This is a single centre, single arm, preoperative window of opportunity study with a biomarker endpoint (expression profiling by RNA sequencing). Patients with resectable, histologically confirmed head and neck squamous cell carcinoma (HNSCC) for whom surgical treatment is planned as definitive management will be eligible. The median time from consultation to major head and neck surgery at our institution is 3.2 +/- 2.0 weeks (1 standard deviation). To provide the maximal opportunity to achieve a biomarker response and potentially observe clinical responses, patients will receive BYL719 orally daily at the maximum tolerated dose (400 mg/day) for 14 days. All patients will receive surgery as the standard of care. The gene expression profile, including Ki-67, from the surgical specimen and mandatory baseline tumor biopsy will be evaluated for primary and secondary pharmacodynamic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed squamous cell carcinoma of the head and neck.
* Patients must be eligible for curative intent treatment with surgical resection
* Patients have measurable disease measuring 10 mm or more by clinical exam using calipers according to RECIST 1.1 criteria. Caliper examination must be within 1 week of registration.
* Patients are able to swallow and maintain oral medication
* Prior systemic therapy and/or radiotherapy are allowed if therapy was completed ≥12 weeks prior to BYL719 treatment start date.
* Age ≥18 years.
* Ability to understand and the willingness to sign a written informed consent document and is able to comply with protocol requirements.
* ECOG performance status ≤ 2 (Karnofsky ≥60%). See Appendix A.
* Life expectancy of greater than 6 months.
* Patients must have adequate organ and marrow function done within 2 weeks of starting treatment as defined below:

  1. Leukocytes ≥ 3.0 x 109/L
  2. Hemoglobin > 90 g/L
  3. absolute neutrophil count ≥1.5 x 109/L
  4. platelets ≥ 100 x 109/L
  5. total bilirubin ≤ 1.5 x institutional upper limit of normal
  6. AST(SGOT) and ALT(SGPT) ≤ 2.5 x institutional upper limit of normal
  7. creatinine ≤ 1.5 x institutional upper limit of normal Or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  8. INR ≤ 1.5
  9. Random plasma glucose ≤ 200 mg/dl or ≤ 11.1 mmol/L
* Women of child-bearing potential must have a negative pregnancy test at screening and agree to use a highly effective method of contraception (IUD or barrier method of birth control or abstinence) during dosing and for 8 weeks after the final dose of study treatment. Hormonal contraceptives may be affected by cytochrome P450 and are therefore not considered effective for this study.
* Males must use a condom during intercourse while taking the study drug and for 4 weeks after the final dose of study medication. In addition to avoiding potential risks to a child conceived while on the study medication, a condom use will prevent delivery of the study drug via seminal fluid.
* Study investigator has reviewed the patient's medication list and has taken appropriate measures if the patient is taking any of the following:

  1. Drugs known to be moderate or strong inhibitors or inducers of isoenzymes CYP34A or CYP2C8
  2. Drugs that are metabolized by CYP450 (CYP3A4, CYP3A5, CYP2C9 and CYP2C19)
  3. BCRP inhibitors
  4. Drugs that may alter gastrointestinal tract pH.
  5. Medications with a known risk of prolonging QT interval or inducing Torsades de Points (TdP)
  6. Warfarin and coumadin derivates
  7. Herbal medications

Exclusion Criteria:

* Patients with known distant metastatic disease
* Patients who have previously received BYL719 or have received any other investigational agents within 30 days.
* Patients with diabetes mellitus requiring insulin or documented steroid induced diabetes mellitus
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (eg. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* History of another malignancy within 2 years prior to starting study treatment, except for cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient has history of hypersensitivity to any drugs or metabolites or similar chemical classes as BYL719
* Patient is currently receiving or has received systemic corticosteroids < 2 weeks prior to starting treatment with BYL719, or has not fully recovered from side effects of such treatment
* Patients who are currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzymes CYP34A or CYP2C8. The patient must have discontinued all such drugs at least 1 week before the start of study treatment. Switching to a different medication prior to treatment start is allowed. Refer to Appendix B for a list of strong and moderate CYP34A and CYP2CA inducers and inhibitors.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information

* Patient receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot be discontinued or switched to a different medication prior to starting study treatment. Refer to Appendix B, Table 2.
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Patients who have received live attenuated vaccines within 1 week of start of study medication and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Uncontrolled intercurrent illness or medical conditions that would, in the treating physician's judgment, contraindicate patient participation including, but not limited to: active or uncontrolled infection, chronic active hepatitis, immune-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
* Patient has any of the following cardiac abnormalities:

  1. History of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy
  2. known Left Ventricular Ejection Fraction (LVEF) < 50%
  3. myocardial infarction < 6 months prior to enrollment
  4. unstable angina pectoris
  5. serious uncontrolled cardiac arrhythmia
  6. symptomatic pericarditis
  7. QTcF > 480 msec on the screening ECG (using the QTCF formula)
* Patients with known positive serology for human immunodeficiency virus (HIV). HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with BYL719. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patient who has not recovered to grade 1 or better (except alopecia, chronic stable neuropathy or hearing impairment) from related side effects of any prior antineoplastic therapy
* Patient who has undergone major surgery within 14 days prior to starting study treatment or who has not recovered from side effects of such procedure.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL). Patients with elevated hCG at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated 5-7 days later, or pregnancy has been ruled out by vaginal ultrasound.
* Patient who does not apply highly effective contraception during the treatment with BYL719 and through the duration as defined below after the final dose of BYL719:

  1. Sexually active males should use a condom during intercourse while taking drug and for 4 weeks* after the final dose of alpelisib and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
  2. Women of child-bearing potential, defined as all female physiologically capable of becoming pregnant, must use highly effective contraception during the IPP and through at least 4 weeks* after the final dose of alpelisib
  3. Highly effective contraception is defined as either:

  i. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

ii. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before starting treatment with alpelisib. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female patients participating to this IPP, the vasectomized male partner should be the sole partner for that patient] iv. Use a combination of the following (both a+b):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
2. Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as alpelisib BYL719 may decrease the effectiveness of hormonal contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Phospho-S6 (235/6) Expression | Measured at baseline and at surgery
  Phospho-S6 (235/6) measured at baseline from the biopsy tissue sample will be compared to the value measured following BYL719 treatment taken from the tissue removed at surgery using a paired t-test.

SECONDARY OUTCOMES:
Phospho-AKT Levels (Ser473) | Measured at baseline and at surgery
  For Phospho-AKT levels (Ser473) values measured at baseline from the biopsy tissue sample will be compared to the value measured following BYL719 treatment taken from the tissue removed at surgery using a paired t-test.
Ki-67 Levels | Measured at baseline and at surgery
  Ki-67 levels values measured at baseline from the biopsy tissue sample will be compared to the value measured following BYL719 treatment taken from the tissue removed at surgery using a paired t-test.
Severity of Adverse Events | At baseline and within 14 days of last dose
  The frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious, and severe events of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Nichols, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London Regional Cancer Program, London, Ontario, Canada

REFERENCES:
- [Derived] Ruicci KM, Meens J, Sun RX, Rizzo G, Pinto N, Yoo J, Fung K, MacNeil D, Mymryk JS, Barrett JW, Boutros PC, Ailles L, Nichols AC. A controlled trial of HNSCC patient-derived xenografts reveals broad efficacy of PI3Kalpha inhibition in controlling tumor growth. Int J Cancer. 2019 Oct 15;145(8):2100-2106. doi: 10.1002/ijc.32009. Epub 2018 Dec 18. PMID 30468243